CLINICAL TRIAL: NCT04371263
Title: How Dose Election Event Will Induce Emotion Change of Emergency Room and Critical Unit and What is the Influence of Emotional Change in the Daily Duty
Brief Title: How Dose Election Event Will Induce Emotion Change of Emergency Room and Critical Unit
Status: Completed | Type: Observational
Sponsor: St. Martin De Porress Hospital (Other)
Responsible Party: Principal Investigator, Chia-hsi Chen, Attending Physician of Emergency Department, St. Martin De Porress Hospital
Other Study IDs: 19B-003
Record Dates: First submitted 2020-03-24; First posted 2020-05-01 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Emotional Problem
Keywords: emotional change; emotional labor; emotional control
MeSH Terms: interventions — Emergency Service, Hospital

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Emotional Change of Nursing Manpower in Emergency and Critical Unit After Keen Election And What's The Influence of Emotional Change — use the emotion regulation questionnaire (ERQ) to realize the influence in duty work

SUMMARY:
In response to the emergence of injuries and illnesses, the manpower of the acute and critical medical team has the requirements. The election keen is rare to see in recent years. The results of the election event will inevitably bring to the emergency and critical unit nursing staff and on-site counter personnel. Certain emotional changes is noted and this study is to understand the impact of the emotional adjustment of personnel in acute and critical units on their own work, to understand the situation of on-site personnel, and to avoid excessive planning of manpower, which will help hospital manpower deployment

I

DETAILED DESCRIPTION:
In 20181124, the mayor of the county and the 2020 president election, after the election, the mood changes of the nursing staff of the emergency and critical unit and the staff of the on-site counter medical department were filled out with a questionnaire to understand the mood changes of the nursing staff and on-site counter staff in each unit and how to adjust Analysis of the impact on clinical work. Exclude those who complete the questionnaire data incompletely, the statistical method used is to calculate the Cronbach's α and correlation coefficient for the questionnaire sample verification.

ELIGIBILITY:
Inclusion Criteria:

* Nursing Manpower in Emergency and Critical Unit

Exclusion Criteria:

* Incomplete questionnaire filled in

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Nursing Manpower in Emergency and Critical Unit
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2018-11-24 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
The Emotional Change of Nursing Manpower in Emergency and Critical Unit After Keen Election Impaction And What's The Influence of Emotional Change | through study completion, an average of 1 and half year
  emotional change will has influence in nursing care activity after the knee election. One questionnaire such as EMOTION REGULATION QUESTIONNAIRE is used in The emotional control survey.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Martin De Porres Hospital, Chiayi City, Taiwan